CLINICAL TRIAL: NCT00232804
Title: Safety and Efficacy Registry of Bx Cypher Stent in the Revascularisation of Patients With Significant Risk of Restenosis
Brief Title: The BRIDGE Registry: Safety and Efficacy Registry of Bx Cypher Stent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01290402
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Device: Bx Cypher stent

INTERVENTIONS:
Device: Bx Cypher stent

SUMMARY:
The objective of this study is to establish the safety and efficacy of the treatment with Cypher DES in diabetic patients with documented ischemia due to stenosis (small coronary artery 2.5 -3 mm in lumen diameter, with lesion between 15 mm 30 mm in length, ) in native coronary arteries.

The objective of this study is to document that the use of Cypher DES in these diabetic patients undergoing percutaneous revascularization for stenosis is safe.

Safety will be assessed over a period of 12 months.

DETAILED DESCRIPTION:
This is a prospective, multicenter, comparative, non randomised, open registry of 1000 patients who will be followed up to 12 months at 100 sites in France.

Patients will be screened according to normal practice and in relation to the inclusion and exclusion criteria. Patients should have a documented ischemia related to the target vessel.

Procedure of stent placement should be done under existing in hospital procedural protocol and care should be taken to follow Cordis instructions as set forth in the Instructions For Use.

Follow up will be done according to normal procedure and the minimum should be a telephone contact at 1, 6 and 12 months.

All data gathered during the enrollment, procedure, follow up and when specific events to the patient may occur, will be entered into the Internet CRF form, by the treating physician or a person from his staff specifically appointed to this task.

Patient enrollment is anticipated to last 8 months.

ELIGIBILITY:
Inclusion Criteria:

1. NIDDM treated with oral antidiabetics for at least 3 months, or IDDM treated for at least 3 months with documented HbA1C;
2. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B I-II) OR patients with documented silent ischemia;
3. Target lesion stenosis is >50% (visual estimate);
4. Target vessel diameter, between 2.5 and 3.0 mm
5. Target lesion length minimum 15 mm and maximum 30mm

Exclusion Criteria:

1. CK and CK-MB enzymes above normal or elevated troponin level (as determined by site criteria) at the time of treatment;
2. Has unstable angina classified as Braunwald III B and A or C I-II-III, or is having a peri-infarction;
3. Unprotected left main coronary disease with >=50% stenosis;
4. Significant (>50%) stenosis proximal or distal to the target lesion that might impede inflow or runoff and can not be revascularized before or during the index procedure;
5. Have an ostial target lesion;
6. Documented left ventricular ejection fraction <=30%;
7. In-Stent restenosis;
8. Chronic total occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2002-06; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
MACE. | 1, 6, and 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lablanche, Prof., Principal Investigator — Université de Lille, Hôpital cardiologique
Locations (1):
- Université de Lille, Hôpital cardiologique, Lille, France

REFERENCES:
- [Result] Lablanche JM, Commeau P; Investigateurs du Registre BRIDGE. [BRIDGE registry (safety and efficacy registry Bx Cyper stent in the RevascularIzation of patients with siGnificative risk of rEstenosis): protocol description and preliminary results]. Ann Cardiol Angeiol (Paris). 2004 May;53 Suppl 1:29s-31s. doi: 10.1016/s0003-3928(04)90006-6. No abstract available. French. PMID 15291158